CLINICAL TRIAL: NCT03224923
Title: Reassessment of Long-Term Dual Anti-Platelet Therapy Using InDividualized Strategies - Using a Novel Combined Demographic and Pharmacogenomic Strategy: The RAPID EXTEND Pilot Study
Brief Title: A Novel Strategy For Personalized Long-Term Dual Antiplatelet Therapy (RAPID EXTEND PILOT STUDY)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Competing study to be started in November 2018
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170341
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Stable Coronary Syndrome; Percutaneous Coronary Intervention; Antiplatelet Therapy; Ticagrelor
MeSH Terms: interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Treatment Algorithm (Experimental): A DAPT score using various patient demographics will be calculated:
  If score under 2, patients will receive only aspirin 81 mg once daily
  If DAPT score is ≥ 2
  * A point-of-care bedside genetic test using a buccal swab will be conducted in order to determine medication regimen
  * Those with a positive genetic test (presence of CYP2C19*2 or CYP2C19*3), will receive 60mg Ticagrelor twice daily
  * Those with a negative genetic test (absence of CYP2C19*2/*3) will receive 75mg clopidogrel once daily
  Interventions: Drug: Ticagrelor 60mg; Drug: Clopidogrel 75mg; Drug: Aspirin 81 mg
- Long-Term Ticagrelor (Active Comparator): Patients will be given 60mg Ticagrelor twice daily with no aspirin
  Interventions: Drug: Ticagrelor 60mg

INTERVENTIONS:
Drug: Ticagrelor 60mg — twice daily
Drug: Clopidogrel 75mg — once daily
  Arms: Personalized Treatment Algorithm
Drug: Aspirin 81 mg — once daily
  Arms: Personalized Treatment Algorithm

SUMMARY:
In patients with heart attacks, the current standard of care is to restore blood flow through percutaneous coronary intervention (PCI). This is done using stents (metal meshes) that opens up blockages. Following PCI, standard preventative drug treatment includes the use of dual antiplatelet therapy (DAPT) using both aspirin and a platelet P2Y12 receptor inhibitor (Ticagrelor 90 mg twice a day or Clopidogrel 75 mg once a day) for one year to prevent clotting that can result in additional heart attacks, sudden clotting of stents or death.

New studies have shown that there is a benefit to continuing DAPT beyond this one year mark. Longer-term DAPT has been shown to reduce ischemic events (heart attack, stroke) but increase the risk of bleeding. Present guidelines state that the decision to continue DAPT beyond the one year mark should be made on an individualized basis.

The present study is a "pilot study" that seeks to compare Long-Term use of Ticagrelor (LTT) versus a Personalized Approach (PA). We will be recruiting patients who have been stable (free of ischemic or bleeding outcomes) on DAPT for 1 year after initial presentation with a heart attack.

The PA group will use a modified DAPT score based on patient demographics to decide whether treatment is warranted. Patient will also undergo bedside genetic testing to identify potential at-risk genes. Those identified as carriers will be treated with ticagrelor while non-carriers will be treated with clopidogrel.

The present study will determine whether a personalized approach will decrease bleeding versus an approach of universal ticagrelor use.

The hypothesis is that patients receiving a personalized strategy will have a decreased risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* non-ST-elevation myocardial infarction (NSTEMI) or ST-elevation myocardial infarction (STEMI) at presentation for index PCI who have successfully completed >1-year follow-up of RAPID MANAGE or TAILOR-PCI trials without having incurred an ischemic or bleeding outcome while on DAPT
* Patients with DAPT interruption after 1 year will be eligible, if within 3 years of index MI

Patients must also have 1 of the following atherothrombotic risk enrichment criteria:

* age ≥ 65 years
* diabetes
* 2nd prior MI (> 1 year ago)
* multi-vessel coronary disease
* Creatinine Clearance < 60mL/min

Exclusion Criteria:

Patients will be excluded from the study if they:

* refuse consent
* are > 3 years post MI
* are deemed to require a P2Y12 inhibitor
* require oral anticoagulation
* have a history of stroke, transient ischemic attack (TIA) or intracranial bleed
* have had a recent GI bleed or major surgery
* have a life expectancy of < 1 year
* have a platelet count < 100,000/μl
* have a bleeding diathesis
* have hematocrit < 30% or > 52%
* are on dialysis or have severe liver disease
* are at risk for bradycardia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with Decreased Bleeding Risk | 1 month
  The primary endpoint is the proportion of patients with low on-treatment platelet reactivity (LPR) in the PA group compared to the LTT group at 1 month.
  * P2Y12 reactivity units (PRU) as a continuous variable will be measured using a VerifyNow P2Y12 assay
  * a PRU value of < 85 is associated with increased bleeding risk

SECONDARY OUTCOMES:
Platelet Reactivity Index (PRI) as a continuous variable | 1 month
  Platelet function as measured by Vasodilator-stimulated phosphoprotein (VASP)
  * a PRI of < 16% is associated with increased bleeding risk
ADP-induced Aggregation (AU) as a continuous variable | 1 month
  Platelet function as measured by Multiplate analyzer
  * an AU of < 19 is associated with increased bleeding risk
Bleeding according to Bleeding Academic Research Consortium (BARC) criteria | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  the incidence and severity of bleeding as defined by BARC classification system
Bleeding according to Thrombolysis in Myocardial Infarction (TIMI) score | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  the incidence and severity of bleeding as defined by TIMI classification systems
Bleeding according to Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO) criteria | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  the incidence and severity of bleeding as defined by GUSTO classification systems
Ischemic Endpoints (To be collected but blinded to investigators, as this data will be carried from the pilot study into a future definitive clinical trial). | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  all-cause mortality incidence
Ischemic Endpoints (To be collected but blinded to investigators, as this data will be carried from the pilot study into a future definitive clinical trial). | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  recurrent myocardial infarction (MI) incidence
Ischemic Endpoints (To be collected but blinded to investigators, as this data will be carried from the pilot study into a future definitive clinical trial). | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  stroke incidence
Ischemic Endpoints (To be collected but blinded to investigators, as this data will be carried from the pilot study into a future definitive clinical trial). | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  stent thrombosis incidence

OTHER OUTCOMES:
Cost | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  Evaluate cost involved in each strategy
Genetic factors associated to outcomes | 1 month, 6 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years
  Exploratory analysis of other potential genetic variants to outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Derek So, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada